CLINICAL TRIAL: NCT00217217
Title: Low Field Magnetic Stimulation in Bipolar Depression
Brief Title: Low Field Magnetic Stimulation Treatment for Bipolar Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated for lack of recruitment.
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2004P-002631
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Depression; Bipolar Disorder; Depression
Keywords: non-pharmaceutical; alternative; imaging; magnetic resonance imaging; low field magnetic stimulation; bipolar disorder; depression; bipolar depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Echo-Planar Imaging

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active EEP-MRSI treatment (Experimental): 20 minutes of active treatment with theEcho-Planar Magnetic Resonance Imaging (EP-MRSI)
  Interventions: Device: Echo-Planar Magnetic Resonance Imaging (EP-MRSI)
- Sham comparator EP-MRSI (Sham Comparator): Sham treatment (20 minutes) with the Echo-Planar Magnetic Resonance Imaging (EP-MRSI).
  Interventions: Device: Echo-Planar Magnetic Resonance Imaging (EP-MRSI)

INTERVENTIONS:
Device: Echo-Planar Magnetic Resonance Imaging (EP-MRSI) — variable-setting low-frequency MRI
  Other Names: Low Field Magnetic Stimulation (LFMS)

SUMMARY:
Individuals with bipolar depression who had a particular kind of brain imaging reported improved mood after the imaging. This effect may be linked to the changing magnetic fields used during these magnetic resonance imaging studies. The current studies are designed to further explore the important parameters of this effect and to clarify the degree and duration of the mood effects.

DETAILED DESCRIPTION:
An initial study using proton echo-planar magnetic resonance spectroscopic imaging (EP-MRSI) in bipolar depressed individuals was associated with reports of improved mood. These studies employed oscillating magnetic fields similar to those used in functional MRI (fMRI), but which differ from the usual fMRI scan in field direction, waveform frequency, and strength. As the abbreviation EP-MRSI is used to describe several relatively common MR sequences, the specific potential clinical procedure being used is referred to as low field magnetic stimulation or LFMS. Following these initial results, investigators are conducting studies to determine the critical variables in both subjects and treatment for optimal response. Studies are also underway to characterize the response of specific depression symptoms, the degree of response, and the duration of response.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of bipolar disorder.
* Current depression.

Exclusion Criteria:

* Contraindication for MRI due to metal in eyes/head
* Claustrophobia.
* Inability to lie flat.
* History of brain injury.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Scale | pre/post-treatment

SECONDARY OUTCOMES:
Visual-Analog Scales | pre/post-treatment
Montgomery Asberg Depression Rating Scale (MADRS) | pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rohan, MS, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Carlezon WA Jr, Rohan ML, Mague SD, Meloni EG, Parsegian A, Cayetano K, Tomasiewicz HC, Rouse ED, Cohen BM, Renshaw PF. Antidepressant-like effects of cranial stimulation within a low-energy magnetic field in rats. Biol Psychiatry. 2005 Mar 15;57(6):571-6. doi: 10.1016/j.biopsych.2004.12.011. PMID 15780843
- [Result] Rohan M, Parow A, Stoll AL, Demopulos C, Friedman S, Dager S, Hennen J, Cohen BM, Renshaw PF. Low-field magnetic stimulation in bipolar depression using an MRI-based stimulator. Am J Psychiatry. 2004 Jan;161(1):93-8. doi: 10.1176/appi.ajp.161.1.93. PMID 14702256